CLINICAL TRIAL: NCT02420379
Title: An Open-Label, Multi-Center Study to Evaluate the Safety, Efficacy and Tolerability of Eteplirsen in Early Stage Duchenne Muscular Dystrophy
Brief Title: Safety Study of Eteplirsen to Treat Early Stage Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4658-203
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: DMD; Duchenne muscular dystrophy; eteplirsen; Dystrophin; exon 51
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-Label (Experimental): Approximately 20 patients will receive weekly infusions of eteplirsen 30 mg/kg .
  Interventions: Drug: eteplirsen
- Control Group (No Intervention): Approximately 20 patients with DMD not amenable to exon 51 skipping will be observed for 96 weeks.

INTERVENTIONS:
Drug: eteplirsen — Eteplirsen 30 mg/kg will be administered as an IV infusion once a week for 96 weeks.
  Other Names: AVI-4658; EXONDYS 51®
  Arms: Open-Label

SUMMARY:
This is an open-label study to assess the safety, tolerability, efficacy and pharmacokinetics of eteplirsen in patients with early stage Duchenne muscular dystrophy (DMD) who are amenable to exon 51 skipping.

DETAILED DESCRIPTION:
Safety, including adverse event monitoring and routine laboratory assessments, will be followed on an ongoing basis for all patients.

Clinical efficacy, including functional tests and MRI, will be assessed at regularly scheduled study visits. Patients will undergo one baseline and one follow-up muscle biopsy.

Population and serial PK will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male 4-6 years of age.
* Diagnosis of DMD, genotypically confirmed.
* Stable dose of oral corticosteroids for at least 12 weeks or has not received corticosteroids for at least 12 weeks.
* Intact right and left biceps muscles or two alternative upper arm muscle groups.
* Parent that is willing to provide consent and comply with study procedures.

Exclusion Criteria:

* Use of any pharmacologic treatment (other than corticosteroids) within 12 weeks that may have an effect on muscle strength or function (e.g., growth hormone, anabolic steroids).
* Previous or current treatment with any other experimental treatments within 12 weeks or participation in any other clinical trial within 6 months.
* Major surgery within 3 months prior to the first dose of study drug, or planned surgery during this study which would interfere with the ability to perform study activities.
* Presence of other clinically significant illness.

Ages: 4 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (13):
- United States (13):
  - Neuromuscular Research Center of Arizona, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Rare Disease Research Center, Atlanta, Georgia
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 sites in the United States.
Pre-assignment Details: A total of 33 participants were enrolled in the study treatment.
Groups:
- Eteplirsen 30 mg/kg: Participants with Duchenne muscular dystrophy (DMD) amenable to exon 51 skipping received eteplirsen 30 milligram per kilogram (mg/kg) intravenous (IV) infusions, once weekly, for 96 weeks.
- Control Group (Untreated) (Non-exon 51 Amenable Participants): Participants with DMD not amenable to exon 51 skipping were observed for 96 weeks.
Period: Overall Study
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Started | 26 | 7
Completed | 25 | 3
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Unable to complete due to schooling | 0 | 1
Not completed — Transitioned to commercial drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full set included all participants who were enrolled in the eteplirsen group and received at least 1 dose of eteplirsen as well as all participants who were enrolled in the untreated group and had at least 1 assessment post-enrollment assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants) | Total
Number analyzed (Participants) | 26 | 7 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (0.82) | 5.0 (1.00) | 5.0 (0.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 7 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 21 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 6 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: Adverse Event (AE) was any untoward medical occurrence in a participant that did not necessarily have a causal relationship with the study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; Life-threatening event; required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Treatment emergent adverse events were events that developed or worsened during the on-treatment period (defined as time from first dose of study drug and up to 28 days after last dose of study drug [up to 100 weeks]) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 100 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants
  Participants with TEAEs | 26 | 5
  Participants with Serious TEAEs | 4 | 0
  Participants with TEAEs leading to discontinuation | 0 | 0

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities Reported as TEAEs
Description: Laboratory parameters included hematology, serum chemistry (SC), urinalysis and coagulation. Number of participants with at least one potentially clinically significant abnormal findings were reported as TEAEs. The Investigator determined whether abnormal assessment results were clinically significant or not clinically significant. Clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to 100 weeks
Population: Full set included all participants who are enrolled in the eteplirsen group and receive at least 1 dose of eteplirsen as well as all participants who are enrolled in the untreated group who have at least 1 assessment post-enrollment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants
  SC: Blood creatine phosphokinase increased | 1 | 0
  Hematology: Anaemia | 1 | 0
  Hematology: Iron deficiency Anaemia | 1 | 0
  Urinalysis: chromaturia | 3 | 0
  Urinalysis: pollakiuria | 1 | 0
  Coagulation: Thrombocytopenia | 0 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs Reported as TEAEs
Description: Vital sign parameters included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and body temperature. Number of participants with at least one potentially clinically significant abnormal vital signs findings were reported as TEAEs. The Investigator determined whether abnormal assessment results were clinically significant or not clinically significant. Clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to 100 weeks
Population: Full set included all participants who were enrolled in the eteplirsen group and receive at least 1 dose of eteplirsen as well as all participants who are enrolled in the untreated group who have at least 1 assessment post-enrollment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants
  Pyrexia | 11 | 1
  Pulse pressure increased | 1 | 0
  Tachycardia | 1 | 0

4. Primary Outcome: Number of Participants With at Least One Abnormal Physical Examination Finding
Description: Physical examinations, full and brief, were performed by the Investigator, a physician Sub-Investigator, or a Nurse Practitioner (if licensed in the state or province to perform physical examinations). Full physical examinations included examination of general appearance; head, ears, eyes, nose, and throat; heart; lungs; chest; abdomen; skin; lymph nodes; and musculoskeletal and neurological systems. Number of participants with at least one abnormal physical examination findings were reported. Abnormality in physical examinations was based on Investigator's discretion.
Time Frame: Baseline up to 100 weeks
Population: Full set included all participants who are enrolled in the eteplirsen group and receive at least 1 dose of eteplirsen as well as all participants who are enrolled in the untreated group who have at least 1 assessment postenrollment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants | 23 | 4

5. Primary Outcome: Number of Participants With Abnormalities in Electrocardiograms (ECGs) Reported as TEAEs
Description: Twelve-lead ECGs and Holter ECGs were performed at a consistent time of day throughout the study. Electrocardiograms were performed only after the participant was in the supine position, resting, and quiet for a minimum of 15 minutes. The ECG was manually reviewed and interpreted by medically qualified personnel. Number of participants with at least one abnormalities in ECGs were reported as TEAEs.
Time Frame: Baseline up to 96 weeks
Population: Full set included all participants who are enrolled in the eteplirsen group and receive at least 1 dose of eteplirsen as well as all participants who are enrolled in the untreated group who have at 1 assessment post-enrollment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants | 1 | 0

6. Primary Outcome: Number of Participants With Abnormalities in Echocardiograms (ECHO) Reported as TEAEs
Description: Standard, 2-dimensional ECHOs were performed at a consistent time of day throughout the study. Cardiac function events included cardiomegaly, tachycardia, and dyspnoea. The ECHO was reviewed and interpreted by medically qualified personnel. Number of participants with at least one abnormalities in ECHO were reported as TEAEs.
Time Frame: Baseline up to 96 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
Number analyzed (Participants) | 26 | 7
Participants | 1 | 0

7. Secondary Outcome: Change From Baseline in Dystrophin Protein Levels Quantified by Western Blot at Week 48 and 96
Description: Change from baseline in dystrophin protein levels (in muscle biopsy samples) were determined by Western blot at Week 48 and 96 was reported. For each time point, 2 blocks of tissues were analyzed by Western blot, each with 2 replicates of gels to determine the dystrophin level as compared to a healthy individual (Percent Normal). The block average value from 2 replicate gels was computed. The overall average was calculated as the mean of the block average values. The overall average values were used for all analyses. In case only 1 gel was available for a block, then that value was used as the block average value.
Time Frame: Baseline, Week 48 and 96
Population: Muscle Biopsy Set included all participants who received at least 1 dose of eteplirsen and who had data from both baseline (pre-treatment) and Week 48 or 96 (on-treatment) muscle biopsy samples. Data for this outcome was not planned to be collected and analyzed for control group (untreated) (non-exon 51 amenable participants). Here, number of participants analyzed signifies participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: Percent Normal Dystrophin Protein Level
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 25
Percent Normal Dystrophin Protein Level
  Change at Week 48: number analyzed (Participants) | 14
  Change at Week 48 | 0.102 (0.0896)
  Change at Week 96: number analyzed (Participants) | 11
  Change at Week 96 | 0.321 (0.4863)

8. Secondary Outcome: Change From Baseline in Dystrophin Intensity Levels Determined by Immunohistochemistry (IHC) at Week 48 and 96
Description: Change from baseline in dystrophin intensity levels (in muscle biopsy samples) was determined by Immunohistochemistry at Week 48 and 96 was reported.
Time Frame: Baseline, Week 48 and 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent dystrophin positive fibers
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 25
Percent dystrophin positive fibers
  Change at Week 48: number analyzed (Participants) | 14
  Change at Week 48 | 0.004 (0.0096)
  Change at Week 96: number analyzed (Participants) | 11
  Change at Week 96 | 0.015 (0.0175)

ADVERSE EVENTS:
Time Frame: Baseline up to 100 weeks
Arm/Group | Eteplirsen 30 mg/kg | Control Group (Untreated) (Non-exon 51 Amenable Participants)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/26 | 0/7
Other Adverse Events (participants affected / at risk) | 26/26 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=26) | Control Group (Untreated) (Non-exon 51 Amenable Participants) (N=7)
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Coxsackie viral infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=26) | Control Group (Untreated) (Non-exon 51 Amenable Participants) (N=7)
Nasopharyngitis (Infections and infestations) | 16 | 2
Upper respiratory tract infection (Infections and infestations) | 11 | 1
Ear infection (Infections and infestations) | 8 | 1
Influenza (Infections and infestations) | 5 | 0
Otitis media (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 3 | 0
Rhinitis (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Impetigo (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 11 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 4 | 0
Scratch (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 13 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Pyrexia (General disorders) | 11 | 1
Catheter site pain (General disorders) | 3 | 0
Catheter site bruise (General disorders) | 2 | 0
Headache (Nervous system disorders) | 10 | 0
Migraine (Nervous system disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 7 | 0
Cardiac murmur (Investigations) | 4 | 0
Aggression (Psychiatric disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenoidectomy (Surgical and medical procedures) | 0 | 1
Myringotomy (Surgical and medical procedures) | 0 | 1
Orchidopexy (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement provides that the PI can only publish the study results with the approval of Sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT02420379/SAP_000.pdf
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02420379/Prot_001.pdf